CLINICAL TRIAL: NCT06759389
Title: The VENTOR Clinical Study - VENTilation and Airway Optimization for Cardiac Arrest Resuscitation
Brief Title: The VENTOR Clinical Study
Acronym: VENTOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CoLabs Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP 1.0
Record Dates: First submitted 2024-12-19; First posted 2025-01-06 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Arrest (CA)
MeSH Terms: conditions — Heart Arrest | interventions — Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Ventor (Experimental): Subjects being treated with Ventor device
  Interventions: Device: Resuscitation (Ventor)

INTERVENTIONS:
Device: Resuscitation (Ventor) — Resuscitation with the Ventor device

SUMMARY:
To evaluate the initial safety and effectiveness of the Ventor Airway System in providing short-term ventilation support in non-breathing subjects during cardiopulmonary resuscitation (CPR) and respiratory arrests.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-75 years, inclusive
2. IHCA (non-traumatic)
3. At least 4 feet in height

Exclusion Criteria:

1. Intubated with an endotracheal tube (ET)
2. Valid do-not-attempt-resuscitation (DNAR) or study opt-out bracelet (including previous enrollment bracelet)
3. LAR or Family member objects to enrollment
4. Obvious signs of irreversible death (rigor mortis, dependent lividity, decapitation, transection, decomposition)
5. Responsive with an intact gag reflex
6. Blunt, penetrating, or burn-related injury, drowning, or electrocution
7. Known upper airway foreign body or mass
8. Lower airway obstruction
9. Dental gap of < 2 cm
10. Ingested caustic substances
11. Medicine Admitting Note's medical history is incomplete or has only been completed by an emergency physician.
12. Known esophageal disease or facial/perforating neck trauma defined as study candidates with the following medical history:

    1. Diseases: (Esophageal Varices, Esophageal Cancer, Esophageal Strictures)
    2. Any patient on the following medications will be excluded: (Oxaliplatin, Leucovorin, Fluorouracil)
    3. Any patient with the following examination findings will be excluded: (Caput medusae, History or evidence of vomiting blood)
13. Known vulnerable subject other Inclusion #3, such as known (e.g.: prisoner, pregnancy, terminal illness, dementia)
14. History of medical, surgical or other conditions that, in the opinion of the investigator, would limit study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Ability to provide oxygenation during CPR | From device insertion through 1 hour.
  As measured through the monitoring of intra-arrest PaO2
Ability to provide ventilation during CPR | From device insertion through 1 hour
  As measured through the monitoring of intra-arrest PaCO2
Ability to provide oxygenation during CPR | From device insertion through 1 hour
  As measured through the monitoring of intra-arrest cerebral oximetry
Number of participants with device-related adverse events | From device insertion through 3 months
  Number and rate of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jignesh Patel, M.D., M.Sc., Principal Investigator — Stony Brook University Hospital
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No